CLINICAL TRIAL: NCT04102488
Title: Simplifying Hand Hygiene Technique: Six Steps and 30 Seconds Versus Six Steps and 15 Seconds Versus Three Steps and 30 Seconds Versus Three Steps and 15 Seconds
Brief Title: Simplifying the World Health Organization (WHO) Protocol for Hand Hygiene: Three Steps and 15 Seconds
Acronym: SIHAG II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019-01518; me19Widmer
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Hand Hygiene
Keywords: reduction of bacterial counts; hand hygiene technique

STUDY DESIGN:
Intervention Model Description: two different hand hygiene techniques (six steps and three steps) and two different application times for hand rub (30 seconds and 15 seconds)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 6-step hygiene technique, application time of 30 seconds (Experimental)
  Interventions: Procedure: Six-step hand hygiene technique with an application time of 30 seconds
- 6-step hygiene technique, application time of 15 seconds (Experimental)
  Interventions: Procedure: Six-step hand hygiene technique with an application time of 15 seconds
- 3-step hygiene technique, application time of 30 seconds (Experimental)
  Interventions: Procedure: Three-step hand hygiene technique with an application time of 30 seconds
- 3-step hygiene technique, application time of 15 seconds (Experimental)
  Interventions: Procedure: Three-step hand hygiene technique with an application time of 15 seconds

INTERVENTIONS:
Procedure: Six-step hand hygiene technique with an application time of 30 seconds — Six-step hand hygiene technique with an application time of 30 seconds
  Arms: 6-step hygiene technique, application time of 30 seconds
Procedure: Six-step hand hygiene technique with an application time of 15 seconds — Six-step hand hygiene technique with an application time of 15 seconds
  Arms: 6-step hygiene technique, application time of 15 seconds
Procedure: Three-step hand hygiene technique with an application time of 30 seconds — Three-step hand hygiene technique with an application time of 30 seconds
  Arms: 3-step hygiene technique, application time of 30 seconds
Procedure: Three-step hand hygiene technique with an application time of 15 seconds — Three-step hand hygiene technique with an application time of 15 seconds
  Arms: 3-step hygiene technique, application time of 15 seconds

SUMMARY:
This study is to investigate that non-inferiority in terms of reduction of bacterial counts will be retained when combining the simpler three-step technique for the use of hand rub with a shorter application time of 15 seconds.

DETAILED DESCRIPTION:
The WHO guideline recommends 30 seconds for application of hand rub, however, mean bacterial reduction after 15 seconds of hand rubbing has been recently shown to be non-inferior and shortening application time to 15 seconds has been suggested to improve the frequency of hand hygiene actions in a neonatal care unit. This study is to investigate that non-inferiority in terms of reduction of bacterial counts will be retained when combining the simpler three-step technique for the use of hand rub with a shorter application time of 15 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Medical students are eligible for participation
* Signed informed consent

Exclusion Criteria:

* No signed informed consent

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change of bacterial counts on hands | 30 minutes
  Change of bacterial counts on hands as determined by the mean logarithmic reduction in bacterial counts after performance of hand hygiene

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Widmer, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland